CLINICAL TRIAL: NCT03374007
Title: With Open, Single/Multiple Dosing and Dose Escalation, Phase I Clinical Trial Scheme to Evaluate Safety, Tolerance and Pharmacokinetic Properties of Genolimzumab Injection
Brief Title: Phase I Clinical Trial in Chinese Patients of Advanced and (or) Recurrent Solid Tumor/Lymphoma
Acronym: GB226
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-001
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumor; Recurrent Solid Tumor; Lymphoma; Recurrent Lymphocyte Depleted Classical Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- GB226 1mg/kg single-dose (Experimental): Geptanolimab, 1mg/kg, i.v., single-dose
  Interventions: Biological: Geptanolimab Injection 1mg/kg
- GB226 3 mg/kg single-dose (Experimental): Geptanolimab, 3mg/kg, i.v., single-dose
  Interventions: Biological: Geptanolimab Injection 3mg/kg
- GB226 10mg/kg single-dose (Experimental): Geptanolimab 10mg/kg, i.v., single-dose
  Interventions: Biological: Geptanolimab Injection 10mg/kg
- GB226 1mg/kg multiple dosing, every 2 weeks (Experimental): Geptanolimab, 1mg/kg, i.v., q2w*6
  Interventions: Biological: Geptanolimab Injection 1mg/kg, q2w*6
- GB226 3mg/kg multiple dosing,every 2 weeks (Experimental): Geptanolimab, 3mg/kg, i.v., q2w*6
  Interventions: Biological: Geptanolimab Injection 3mg/kg, q2w*6
- GB226 10mg/kg multiple dosing, every 2 weeks (Experimental): Geptanolimab,10mg/kg, i.v., q2w*6
  Interventions: Biological: Geptanolimab Injection 10mg/kg, , q2w*6
- GB226 280mg multiple dosing (Experimental): Geptanolimab, 280mg, i.v., q3w
  Interventions: Biological: Geptanolimab Injection 280mg, q3w
- GB226 3mg/kg multiple dosing (Experimental): Geptanolimab, 3mg/kg, i.v., q2w
  Interventions: Biological: Geptanolimab Injection 3mg/kg, q2w

INTERVENTIONS:
Biological: Geptanolimab Injection 1mg/kg — single-dose:1mg/kg
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 1mg/kg single-dose
Biological: Geptanolimab Injection 3mg/kg — single-dose: 3mg/kg
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 3 mg/kg single-dose
Biological: Geptanolimab Injection 10mg/kg — single-dose:10mg/kg
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 10mg/kg single-dose
Biological: Geptanolimab Injection 1mg/kg, q2w*6 — multiple dosing: 1mg/kg, q2w*6
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 1mg/kg multiple dosing, every 2 weeks
Biological: Geptanolimab Injection 3mg/kg, q2w*6 — multiple dosing: 3mg/kg, q2w*6
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 3mg/kg multiple dosing,every 2 weeks
Biological: Geptanolimab Injection 10mg/kg, , q2w*6 — multiple dosing: 10mg/kg, , q2w*6
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 10mg/kg multiple dosing, every 2 weeks
Biological: Geptanolimab Injection 280mg, q3w — multiple dosing: 280mg, q3w
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 280mg multiple dosing
Biological: Geptanolimab Injection 3mg/kg, q2w — multiple dosing: 3mg/kg, q2w
  Other Names: Recombinant PD-1 humanized monoclonal antibody injection, Geptanolimab Injection
  Arms: GB226 3mg/kg multiple dosing

SUMMARY:
With open, single/ multiple dosing and dose escalation, phase I clinical trial scheme to evaluate safety, tolerance and pharmacokinetic properties of Genolimzumab injection in Chinese patients of advanced and (or) recurrent solid tumor/lymphoma

DETAILED DESCRIPTION:
Recombinant Programmed death-1(PD-1) humanized monoclonal antibody injection (company code: GB226) is joint developed by Genor Biopharma Co. Ltd and Crown Bioscience,Inc., it is the reorganization of deoxyribonucleic acid (DNA) technology in the Chinese hamster ovary (CHO) cells express system expressed in a immunoglobulin G4 (IgG4) kappa type single resistance to predominate. GB226 had the different new amino acid sequence and molecular structure compared with two marketed PD-1 monoclonal antibody injection and got the approval of China Food and Drug Administration (CFDA) for clinical trial.Pharmaceutical research indicated GB226 cell strain had security source, production process is stable, quality can control, preparation stability, has good compatibility with packaging materials, it has the condition of industrialization, can prepare investigational medicinal product with safety, effective, and controlled quality for clinical research.Pharmacodynamics study show the targets and mechanisms of GB226 is clear, tumor suppression effect is obvious.Toxicology studies show this product in high doses with low toxic, and the toxic is reversible, the most common toxicity is specific to the drug action mechanism.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-65. Unisex.
* 2. Understand trial procedure and content and sign informed consent voluntarily;
* 3. Patients of advanced (phase Ⅲb, multidisciplinary treatment is not appropriate), metastatic (phase IV) or recurrent solid tumor (including melanoma, NSCLC, renal cell carcinoma, head & neck cancer, esophagus cancer, liver cancer, bladder cancer, spongioblastoma) or lymphoma (classical hodgkin lymphoma and (or) peripheral T-cell lymphoma, natural killer (NK)-T cell lymphoma and mediastinal B cell lymphoma) conformed by histology or cytology and cannot be cured by surgery. There is no effective standard treatment now.
* 4. Agree to provide recorded tumor tissue sample or fresh tissue sample.
* 5. Eastern Cooperative Oncology Group (ECOG): 0-1;
* 6. Expected life ≥ 3 months;
* 7. With at least one measurable and evaluable tumor (solid tumor is subject to criteria for evaluating efficacy of Immune-Related Response Criteria (irRC)/RECIST and lymphoma is subject to criteria/revised criteria of international working group);
* 8. Chemotherapy of the whole body is completed at least 4 weeks before inclusion.
* 9. Radiotherapy of the whole body and partial palliative radiotherapy are completed at least 4 weeks before inclusion.
* 10. Corticosteroids (prednisone>10mg/d or equivalent) has been stopped at least 2 weeks before inclusion.
* 11. Autotransplantation is completed at least 3 months before inclusion.
* 12. Major surgeries with the need of general anesthesia are completed at least 4 weeks. Surgeries with the need of local anesthesia/epidural anesthesia are completed at least 2 weeks and the subjects have recovered. Skin biopsies with the need of local anesthesia are completed at least 1 hour before inclusion.
* 13. Previous tumor biotherapy (tumor vaccine, cell factor or growth factor for the purpose of tumor control) is completed at least 4 weeks before inclusion;
* 14. Without severe haematological, cardiopulmonary, liver and kidney diseases except protopathic. For patients of solid tumor, hemoglobin≥9g/dl, neutrophile granulocyte≥1.5×109/L, blood platelet≥100×1012/L. For patients of hematologic tumor, hemoglobin≥8g/dl, neutrophile granulocyte≥1.0×109/L, blood platelet≥80×1012/L.
* 15. Serum creatinine≤1.5xUpper Limit Of Normal (ULN) or creatinine clearance rate≥50mL/min and urine protein<2+ in test paper of urine. For patients with urine protein great than or equal to 2+ in test paper of urine, urine shall be collected in 24 hours and urine protein must less than or be equal to 1g.

etc.

Exclusion Criteria:

* 1. Active central nervous system metastasis; If central nervous system (CNS) metastasis of patients can be treated and their symptoms of nervous system can recover to the baseline level (excluding residual signs or symptoms related to CNS treatment) for 2 weeks when they are included, they can participate in the research. Cranial CT or MRI scanning shall be made for the patients 30 days before inclusion.
* 2. Meningeal metastases or meningeal infiltration of tumors;
* 3. Patients with other malignant tumors (excluding cured cervical carcinoma in situ and skin basal cell carcinoma) shall not participate in the research, unless he/she has been fully relieved at least 2 years without the need of other treatment or other treatment is not needed during the research.
* 4. With active, known or suspected autoimmune disease.
* 5. With previous usage of PD-1 antibody, PD-L1 antibody, PD-L2 antibody or cytotoxic T-lymphocyte-associated antigen-4 immunoglobulin (CTLA-4) antibody for treatment (or other antibody for co-stimulation or check point assess of T cells)
* 6.With severe internal medicine diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, active peptic ulcer, active bleeding.
* 7. With active infection.
* 8. With active tuberculosis infection; with active tuberculosis infection in the past.
* 9. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and treponema pallidum antibody (TP-Ab). Positive subjects of HBsAg may not be excluded from patients of liver cancer.
* 10. Complication with the need of immunosuppressive drug or complication with the need of corticosteroids for whole or partial body in the dosage of immunosuppressive action.

etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
adverse event | all adverse events will be recorded from the time the consent form is signed through 30 days following cessation of treatment.
  adverse event
Serious Adverse Event | all serious adverse events will be recorded from the time the consent form is signed through 30 days following cessation of treatment.
  Serious Adverse Event
Dose limiting Toxicity, DLT | Day 1 to Day 28 after first dose
  Dose limiting Toxicity, DLT
Maximum Tolerated Dose, MTD | Day 1 to Day 28 after first dose
  Maximum Tolerated Dose, MTD

SECONDARY OUTCOMES:
AUC 0-t | up to 12 weeks
  AUC 0-t
C max | up to 12 weeks
  C max
AUC 0-∞ | up to 12 weeks
  AUC 0-∞
T max | up to 12 weeks
  T max
Vd | up to 12 weeks
  Vd
Ke | up to 12 weeks
  Ke
t 1/2 | up to 12 weeks
  t 1/2
CL | up to 12 weeks
  CL
Anti-drug antibody, ADA | up to 12 weeks
  Anti-drug antibody, ADA
IFN-γ concentration | up to 12 weeks
  IFN-γ concentration
peripheral blood CD8+PD-1 receptor occupying ratio | up to 12 weeks
  peripheral blood CD8+PD-1 receptor occupying ratio

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.